CLINICAL TRIAL: NCT00668343
Title: Simvastatin in Relapsing Remitting Multiple Sclerosis (RRMS) Patients Using Avonex Compared to Placebo
Acronym: irmsrct
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: mansoureh togha, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132/9388; 83/132/9388
Record Dates: First submitted 2008-04-27; First posted 2008-04-29 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: edss attack
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: simvastatin
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: simvastatin — 40 mg/ day
  Arms: 1
Drug: placebo — 80 mg /day
  Arms: 2

SUMMARY:
Patient with relapsing remitting multiple sclerosis taking avonex are included in this double blind randomized control trial. Simvastatin is compared to placebo. end points of edss , total attack, new enhancing lesion and newt2 lesion in mri is evaluated as end point.

ELIGIBILITY:
Inclusion Criteria:

1. edss<5
2. >=1 attack in last year

Exclusion Criteria:

1. >2 attacks in study
2. drug complication

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
attack number | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mansooreh Togha, MD, Principal Investigator — TUMS
Locations (1):
- Sanaz Ahmadi, Tehran, Iran

REFERENCES:
- [Derived] Togha M, Karvigh SA, Nabavi M, Moghadam NB, Harirchian MH, Sahraian MA, Enzevaei A, Nourian A, Ghanaati H, Firouznia K, Jannati A, Shekiba M. Simvastatin treatment in patients with relapsing-remitting multiple sclerosis receiving interferon beta 1a: a double-blind randomized controlled trial. Mult Scler. 2010 Jul;16(7):848-54. doi: 10.1177/1352458510369147. Epub 2010 May 20. PMID 20488825